CLINICAL TRIAL: NCT07284771
Title: MUSCLE-ML: Multimodal Integration of Muscle Strength, Structure by Machine Learning for Precision Rehabilitation After ACL Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Patrick Shu-Hang YUNG, Professor and Chairman, Department of Orthopaedics & Traumatology, Faculty of Medicine, The Chinese University of Hong Kong, Chinese University of Hong Kong
Other Study IDs: 2025.374; 23241901 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deficit group
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention

SUMMARY:
The goal of this clinical trial is to use machine learning (ML) to predict functional recovery by integrating muscle-related factors and other relevant parameters for identification of non-responders to conventional rehabilitation. The main questions it aims to answer are:

Do deficit clusters lead to poorer functional recovery compared to non-deficit clusters? Does an ML-derived composite score that integrates quadriceps/hamstring strength and size outperform isolated metrics in predicting RTP success?

Researchers will compare deficit clusters against non-deficit clusters to determine if deficit clusters lead to poorer functional recovery.

Participants will:

Return for 5 follow-up timepoints in total for PRO and functional assessments including pre-operation, 1-, 3-, 6- and 12-months post-operation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ACL injury and plan for ACLR
* Commit the post-operation physiotherapy in Prince of Wales Hospital

Exclusion Criteria:

* Preoperative radiographic signs of arthritis
* Patient non-compliance to the rehabilitation program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the ACLR patients will be recruited at the Orthopaedics Outpatient Clinic at Prince of Wales Hospital.
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee score | 6- and 12-months post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Shu Hang YUNG, Principal Investigator — Chinese University of Hong Kong